CLINICAL TRIAL: NCT03744039
Title: Management of Diabetic Patients With Neuropathic Osteoarthropathy (Charcot Foot) : Descriptive Study in Diabetic-foot Centers.
Acronym: EPiChar
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: 30RC18_0078; 2018-A01721-54 (Other: ANSM)
Record Dates: First submitted 2018-11-09; First posted 2018-11-16 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2021-08

CONDITIONS: Diabetic Foot Neuroarthropathy Charcot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite the prominence of diabetes prevalence (more than 8% of the world population in 2012) and its expected increase in the next 15 years, Charcot foot remains a widely unknown diabetes complication. At this day, there is no national guidelines about diagnosis and treatment of this complication, which is known to alter life quality and to increase risk of foot ulceration and mortality in diabetics. Through this descriptive multicentric study, we will investigate the Charcot foot cares in diabetic-foot centers in France and Belgium.

ELIGIBILITY:
Inclusion Criteria:

* The patient has received written information about the study and did not oppose to participate
* The patient is affiliated to a health insurance programme
* The patient is at least 18 years old
* The patient is admitted to hospitalization or consultation
* The patient is diagnosed with type 1 or type 2 diabetes mellitus
* The patient is diagnosed with acute or chronic osteo-neuroarthropathy

Exclusion Criteria:

* The patient participates in another interventional study
* The patient refuses to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 290-1160 consecutive patients with type 1 or type 2 diabetes mellitus and acute or chronic osteo-neuroarthropathy in 29 diabetic-foot centers in France and Belgium (members of workgroup " diabetic foot " in French-speaking Society of Diabetology)
Sampling Method: Non-Probability Sample
Enrollment: 1160 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
Charcot foot's diagnostic criteria | inclusion visit
  triggering factors : yes/no acute symptoms : : yes/no chronic symptoms : yes/no Presence of associated soft tissue infection : yes/no Presence of an associated bone infection : yes/no examinations performed to confirm the diagnosis of Charcot : yes/no
Description Charcot foot's treatment | inclusion visit
  Discharge used in acute phase and/or in case of wound : yes/no Shoes used in chronic phase : yes/no

SECONDARY OUTCOMES:
Number of Charcot foot | inclusion visit
  To determine diabetic patients' number with acute or chronic Charcot foot cared in diabetic-foot center in France and Belgium over a year (estimation of Charcot foot's incidence in diabetic-foot centers).
Surgery of Charcot foot | inclusion visit
  To identify which diabetic-foot centers propose surgical management in Charcot foot, to describe the type of surgery and the indications of surgical treatment.
Register of Charcot foot | inclusion visit
  participation to a register of Charcot foot : yes/no

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de Nîmes - Hôpital Universitaire de Réadaptation du Grau du Roi, Le Grau-du-Roi
  - Nimes University Hospital, Nîmes

REFERENCES:
- [Result] Dardari D, Schuldiner S, Julien CA, Ha Van G, M'Bemba J, Bourgeon M, Sultan A, Lepeut M, Grandperret-Vauthier S, Baudoux F, Francois M, Clavel S, Martini J, Vouillarmet J, Michon P, Moret M, Monnier A, Chingan-Martino V, Rigalleau V, Dumont I, Kessler L, Stifii I, Bouillet B, Bonnin P, Lemoine A, Da Costa Correia E, Faraill MMB, Muller M, Cazaubiel M, Zemmache MZ, Hartemann A. Trends in the relation between hyperglycemia correction and active Charcot neuroarthropathy: results from the EPICHAR study. BMJ Open Diabetes Res Care. 2022 Sep;10(5):e002380. doi: 10.1136/bmjdrc-2021-002380. PMID 36215101